CLINICAL TRIAL: NCT05496049
Title: Efficacy of Triburter on Respiratory Muscle Function in Patients with CABG Who Belong to Cardiac Rehabilitation Phase II Coronary Artery Bypass Graft
Brief Title: Efficacy of Triburter on Respiratory Muscle Function in Patients After CABG in Cardiac Rehabilitation Phase II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI-2022-04334
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Thoracic Surgery; Postoperative Period; Weakness, Muscle
Keywords: Triburter; Respiratory muscle strength; Postoperative patients; Coronary artery bypass graft surgery; Respiratory Therapy
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups by a randomization list provided by a computer program. The intervention group will receive a triburter device for training, the patients will have to repeat 50 ventilations (start with 20 repetitions in the first week, 30 in the second, 40 in the four week, and 50 in the last week) five days per day. For the control group (incentive spirometry) they will repeat 10 ventilations per 5 five times a day. Both interventions will be performed for 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triburter (Experimental): The intervention group will receive a triburter device for training, the patients will have to repeat 50 ventilations (start with 20 repetitions in the first week, 30 in the second, 40 in the four week, and 50 in the last week) five days per day.
  Interventions: Device: Triburter
- Incentive spirometry (Active Comparator): For the control group (incentive spirometry) they will repeat 10 ventilations per 5 five times a day. Both interventions will be performed for 4 weeks.
  Interventions: Device: Incentive spirometry

INTERVENTIONS:
Device: Triburter — Patients will have to repeat 50 ventilations (start with 20 repetitions in the first week, 30 in the second, 40 in the four week, and 50 in the last week) five days per day for four weeks. And they have to fill a calendar to ensurance the intervention.
  Other Names: Triburter device
  Arms: Triburter
Device: Incentive spirometry — They will repeat 10 ventilations per 5 five times a day. Both interventions will be performed for 4 weeks. They have to fill a calendar to ensurance the intervention.
  Arms: Incentive spirometry

SUMMARY:
Post-surgery patients have muscle impairments, especially in the respiratory muscles, because the anesthesia, surgical incision, mechanical ventilation, pain, and prolonged postures, affect the mechanical condition of respiratory muscles. Those consequences produce a low exercise tolerance and low quality of life. These patients must go to cardiac rehabilitation to improve heart functions; however, these patients have a weakness in their respiratory muscles. Currently, there are many devices for respiratory muscle strength, although these devices are expensive, and they only have one circuit for training (inspiratory or expiratory). Triburter is a new device with two valves and positive pressure generation, this is a promising alternative because Triburter improves the mechanics of ventilation, increasing their functionality and quality of life. For this reason, the main hypothesis is that respiratory muscle training with Triburter improves the strength of inspiratory and expiratory muscles.

DETAILED DESCRIPTION:
Aim and objectives: The aim of this study is to determine the efficacy of the Triburter device in comparison with usual therapy (incentive spirometer), as a therapeutic element in respiratory therapy on respiratory muscle function in patients with cardiovascular surgery who will join the second phase of the cardiac rehabilitation program of Fundación Cardiovascular de Colombia. And the specific objectives will be to evaluate the magnitude of change of maximal inspiratory pressure and maximal expiratory pressure, lung function (spirometry), functional capability (6MWT), quality of life (SF-36) and identify the adverse events related to the use of Triburter or incentive Methods design: The design of the pilot study is a randomized clinical trial, open with a control group.

Sample: Following the recommendations to elaborate a pilot trial with feasibility and precision, the recruitment will count 30 patients with no probabilistic sample (intentional sample) Data collection: Personal information forms and case report forms are prepared by principal research after a literature review about relevant variables to collect in the study. CRF included questions regarding socio-economic variables, hospitalized factors, body mass index, heart rate, respiratory rate, and temperature. Then the patients were evaluated in aspects of muscle strength, lung function, functional capacity, and quality of life. The informed consent was obtained from all the patients. The purpose of the study was explained to each patient.

Statistical analyses Firstly, descriptive variables will express in the median and standard deviation for the numeric variables, and for the categoric variables will express in absolute value and percent. A bivariate analysis will be used to determine differences in intergroup through t - Test o Chi-square or U Mann Whitney as appropriate for the type of distribution. The use of crosstabs and categorization of dependent variables to define corresponding patients (with improvement on measures applied) to difference to each group. Correlations will search between clinical variables, functionality, and quality of life through bivariate analysis (spearman) and multivariate (logistic regression) To measure the change induced by training in the functional variables. the researchers will use the analysis of the change of percent [(value pos intervention - value pre/value pre)*100]. To compare the quantitative variables in the two situations (pre-post) and the same group, researchers will use the test of t student for the pair data, and multilevel analysis adjusted by each patient and analyzed by each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients after Coronary Artery Bypass Graft Surgery
* Older 18 years
* Patients that can able to carry out spirometry and volumen lung measures
* Nyha <2
* Patients in phase 2 of cardiac rehabilitation.
* Absent clinical deterioration
* Mechanical ventilation <24 hours after surgery

Exclusion Criteria:

* High risk
* Pneumothorax
* Currently in a clinical trial
* Active smokers
* Patients with COPD
* Major complications hospital period
* Neurological diseases or orthopedic diseases
* Patients who can not be able to carry out the lung function measures.
* Patients with CPAP or BiPAP
* Unable to provide
* Informed consent
* Unstable angina
* Decompensated congestive heart failure.
* Cognitive disorder.
* Uncontrolled arrhythmias.
* Uncontrolled arterial hypertension

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Change in respiratory muscles strength | Day 0, day 14 and day 30
  The maximal inspiratory pressure (cmH2O) and maximal expiratory pressure (cmH2O) allow measure the strength of inspiratory and expiratory muscles. An increase in those pressures means an improvement on respiratory muscle strength

SECONDARY OUTCOMES:
Change in the lung function | Day 0 and day 30
  The lung function will measure by spirometry, specifically the forced expiratory volume in the 1st (Liters) second and forced vital capacity (Liters). An increase in those volumes means an improvement in lung function and expiratory muscles.

OTHER OUTCOMES:
Change in the functional capacity | Day 0 and day 30
  The functional capacity is going to measure by six-minute walk test (meters walking) An increase in meters means an improvement in functionallity.
Change in quality of life | Day 0 and day 30
  The variable quality of life will assess with SF-36 (0-100) with its 6 components( physical function, physic role, body pain, general health, vitality, social function, emotional role and mental health. An increase in these values means an improvement in quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiac Rehabilitation, Piedecuesta, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siafakas NM, Mitrouska I, Bouros D, Georgopoulos D. Surgery and the respiratory muscles. Thorax. 1999 May;54(5):458-65. doi: 10.1136/thx.54.5.458. No abstract available. PMID 10212115
- [Background] Bergofsky EH. Respiratory failure in disorders of the thoracic cage. Am Rev Respir Dis. 1979 Apr;119(4):643-69. doi: 10.1164/arrd.1979.119.4.643. No abstract available. PMID 375788
- [Background] Sobush DC, Dunning M 3rd. Providing resistive breathing exercise to the inspiratory muscles using the PFLEX device. Suggestion from the field. Phys Ther. 1986 Apr;66(4):542-4. doi: 10.1093/ptj/66.4.542. PMID 3960983
- [Background] Restrepo RD, Wettstein R, Wittnebel L, Tracy M. Incentive spirometry: 2011. Respir Care. 2011 Oct;56(10):1600-4. doi: 10.4187/respcare.01471. PMID 22008401
- [Background] Hermes BM, Cardoso DM, Gomes TJ, Santos TD, Vicente MS, Pereira SN, Barbosa VA, Albuquerque IM. Short-term inspiratory muscle training potentiates the benefits of aerobic and resistance training in patients undergoing CABG in phase II cardiac rehabilitation program. Rev Bras Cir Cardiovasc. 2015 Jul-Aug;30(4):474-81. doi: 10.5935/1678-9741.20150043. PMID 27163422
- [Background] Smith JR, Taylor BJ. Inspiratory muscle weakness in cardiovascular diseases: Implications for cardiac rehabilitation. Prog Cardiovasc Dis. 2022 Jan-Feb;70:49-57. doi: 10.1016/j.pcad.2021.10.002. Epub 2021 Oct 22. PMID 34688670
- [Background] Franklin E, Anjum F. Incentive Spirometer and Inspiratory Muscle Training. 2023 Apr 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK572114/ PMID 34283480